CLINICAL TRIAL: NCT03025724
Title: Photodynamic Therapy for Treatment of Cutaneous Squamous Cell Carcinoma in Situ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 897494
Record Dates: First submitted 2016-12-21; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-12

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): After the surgical excision, subjects will be asked to fill out a satisfaction survey. They will not receive any PDT treatment.
- Intervention Group (Experimental): Subjects will undergo a surgical excision of the tumor. Then a clear transparency film will be used to trace the clinical margins of the lesion, as well as any other distinctive skin markings such as nevi or birthmarks. Subjects will then undergo the study procedure where the area to be treated will be swabbed with an alcohol wipe and allowed to dry. Next, the investigator will apply topical 20% 5-ALA (Levulan Kerastick; DUSA Pharmaceuticals) to the SCCis. Then, the area will be occluded with Tegaderm film for 3 hours. At the end of the incubation period, the Tegaderm will be removed and the patient will be exposed to a blue light source (BLU-U; DUSA Pharmaceuticals). Lastly, they will be asked to fill out a satisfaction survey.
  Interventions: Drug: Levulan Kerastick; Device: blue light source; Other: participant satisfaction survey

INTERVENTIONS:
Drug: Levulan Kerastick — Intervention group subjects will undergo a surgical excision of the tumor. Then a clear transparency film will be used to trace the clinical margins of the lesion, as well as any other distinctive skin markings such as nevi or birthmarks. Subjects will then undergo the study procedure where the area to be treated will be swabbed with an alcohol wipe and allowed to dry. Next, the investigator will apply topical 20% 5-ALA (Levulan Kerastick; DUSA Pharmaceuticals) to the SCCis. Then, the area will be occluded with Tegaderm film for 3 hours.
  Other Names: Intervention Group
  Arms: Intervention Group
Device: blue light source — At the end of the incubation period, the Tegaderm will be removed and the patient will be exposed to a blue light source (BLU-U; DUSA Pharmaceuticals).
  Arms: Intervention Group
Other: participant satisfaction survey — Participants will be asked to fill out a satisfaction survey.
  Arms: Intervention Group

SUMMARY:
This pilot study will evaluate the effectiveness of using photodynamic therapy for treatment of cutaneous squamous cell in situ (SCCis). Our hypothesis is that PDT will be effective for treating SCCis. This study will also secondarily evaluate the tolerability of using photodynamic therapy for treatment of SCCis.

Investigators plan to enroll 40 subjects with biopsy proven SCCis. Exclusion criteria include lesion in high-risk site (head, neck, hands, feet), previous severe adverse reaction to topical 20% aminolevulinic acid (Kerastick), previous severe adverse reaction to blue light (BLU-U), allergy to Tegaderm, primary or secondary immunosuppression, history of > 6 skin cancers in the past year, photosensitizing condition such as lupus, or sensitivity to porphyrins.

Age, gender, size, and location of the SCCis will be recorded. All subjects will receive surgical treatment of their SCCis. The control group will undergo a surgical excision of the tumor. After the excision, subjects will be asked to fill out a satisfaction survey. The intervention group will receive PDT plus surgical treatment. Photographs of the lesion will be taken at each study visit. Subjects in the intervention group will then undergo the study procedure of application of topical 20% 5-ALA (Levulan Kerastick; DUSA Pharmaceuticals) to the SCCis. At 3-5 weeks after the initial treatment, the subject will repeat the 3-hour ALA incubation and blue light exposure. At 6 months after the last treatment, subjects in the intervention group will return for clinical follow-up and surgical excision of the lesion. After excision, the specimen will be sent for processing by pathology and subjects will be asked to fill out a satisfaction visual analog scale. All slides will be read by a board-certified dermatopathologist. Side effects will also be monitored using the same graded scale described previously. Mild adverse events that have been associated with PDT, including erythema, skin crusting, superficial blistering, hypopigmentation, and hyperpigmentation. These reactions usually occur during or immediately after the PDT treatment.

DETAILED DESCRIPTION:
Objective: This trial will evaluate the effectiveness of photodynamic therapy (aminolevulinic acid plus blue light) for treatment of cutaneous squamous cell carcinoma in situ (SCCis).

This pilot study will prospectively recruit 40 subjects with biopsy proven SCCis at the time of their visit at University Dermatology East Providence office. Exclusion criteria include lesion in high-risk site (head, neck, hands, feet), previous severe adverse reaction to topical 20% aminolevulinic acid (Kerastick), previous severe adverse reaction to blue light (BLU-U), allergy to Tegaderm, primary or secondary immunosuppression, history of > 6 skin cancers in the past year, photosensitizing condition such as lupus, or sensitivity to porphyrins.

Half of the subjects will be randomized to the control group (n=20), and the remaining subjects (n=20) will be randomized to the intervention group. The subject's age and gender, and size and location of the SCCis will be recorded. For the control group, subjects will undergo a surgical excision of the tumor, which is the gold standard of treatment for SCCis. After the excision, subjects will be asked to fill out a satisfaction survey. They will not receive any PDT treatment.

For the intervention group, photographs of the lesion will be taken at each study visit. A clear transparency film will be used to trace the clinical margins of the lesion, as well as any other distinctive skin markings such as nevi or birthmarks. Subjects will then undergo the study procedure. The area to be treated will be swabbed with an alcohol wipe and allowed to dry. The investigator will apply topical 20% 5-ALA to the SCCis. Then, the area will be covered with Tegaderm film for 3 hours. At the end of 3 hours, the Tegaderm will be removed and the subject will be exposed to a blue light source, which is the standard protocol for treatment with blue light PDT. During administration of the light and immediately afterwards, the subject will be monitored for any side effects, such as erythema, edema, stinging/burning, blisters/crusting, hyperpigmentation, and hypopigmentation. These items will be graded on a scale of 1 to 4 (1=mild and 4=severe) assessed immediately after treatment. This process will be repeated at the next visit 3-5 weeks later. At six months after the last treatment, subjects in the intervention group will return for clinical follow-up and surgical excision of the lesion. Patients will complete a satisfaction survey at the end of this visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18, any gender
2. Biopsy proven SCCis without evidence of microinvasion beyond the epidermis
3. Low-risk site (trunk, arms, legs)
4. Clinical presence of tumor at biopsy site to ensure that biopsy itself was not curative
5. Lesion <2cm
6. Subject amenable to surgical excision at 6 months after the last PDT treatment

Exclusion Criteria:

1. High-risk site (head, neck, hands, feet)
2. Previous severe adverse reaction to topical 20% aminolevulinic acid (Kerastick)
3. Previous severe adverse reaction to blue light (BLU-U)
4. Allergy to Tegaderm
5. Exclusion of any patient with primary or secondary immunosuppression
6. History of > 6 skin cancers in the past year
7. Photosensitizing condition such as lupus
8. Sensitivity to porphyrins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the incidence of SCCis present after exposure to the experimental procedures | six months
  After the excision, investigators will collect patient satisfaction data. Investigators will also review the final pathology report for presence or absence of the tumor.

SECONDARY OUTCOMES:
Physician graded scoring on a 1 to 4 scale of erythema, edema, stinging/burning, blisters/crusting, hyperpigmentation, and hypopigmentation. | six months
  The subjects will be monitored for any side effects, such as erythema, edema, stinging/burning, blisters/crusting, hyperpigmentation, and hypopigmentation. These items will be graded on a scale of 1 to 4 (1=mild and 4=severe) assessed immediately after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kachiu C. Lee, MD, Principal Investigator — University Dermatology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Green A. Changing patterns in incidence of non-melanoma skin cancer. Epithelial Cell Biol. 1992 Jan;1(1):47-51. PMID 1307938
- [Background] Glass AG, Hoover RN. The emerging epidemic of melanoma and squamous cell skin cancer. JAMA. 1989 Oct 20;262(15):2097-100. PMID 2795783
- [Background] Brancaleon L, Moseley H. Laser and non-laser light sources for photodynamic therapy. Lasers Med Sci. 2002;17(3):173-86. doi: 10.1007/s101030200027. PMID 12181632
- [Background] Kennedy JC, Pottier RH, Pross DC. Photodynamic therapy with endogenous protoporphyrin IX: basic principles and present clinical experience. J Photochem Photobiol B. 1990 Jun;6(1-2):143-8. doi: 10.1016/1011-1344(90)85083-9. PMID 2121931
- [Background] Tierney E, Barker A, Ahdout J, Hanke CW, Moy RL, Kouba DJ. Photodynamic therapy for the treatment of cutaneous neoplasia, inflammatory disorders, and photoaging. Dermatol Surg. 2009 May;35(5):725-46. doi: 10.1111/j.1524-4725.2009.01117.x. Epub 2009 Mar 20. PMID 19309338
- [Result] Rogers HW, Weinstock MA, Harris AR, Hinckley MR, Feldman SR, Fleischer AB, Coldiron BM. Incidence estimate of nonmelanoma skin cancer in the United States, 2006. Arch Dermatol. 2010 Mar;146(3):283-7. doi: 10.1001/archdermatol.2010.19. PMID 20231499
- [Result] Miller DL, Weinstock MA. Nonmelanoma skin cancer in the United States: incidence. J Am Acad Dermatol. 1994 May;30(5 Pt 1):774-8. doi: 10.1016/s0190-9622(08)81509-5. PMID 8176018